CLINICAL TRIAL: NCT07052786
Title: Development and Effectiveness Evaluation of a Clustered Care Guideline Within Individualized Developmental Care: RCT
Acronym: Guideline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Fatma Tokan Özkılıçaslan, Lecturer, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/014
Record Dates: First submitted 2025-06-23; First posted 2025-07-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Premature Infant; Clustered Care; Neonatal Intensive Care Unit; Developmental Care
Keywords: clustered care, guideline,nurse, NICU
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (participant blinding) was applied in this study. In order to prevent sample selection bias, the blocks to be used for randomization will be created by a third party
  . The researcher will actively participate in the training and data collection process.
  The ideal method is for the randomization list to be concealed from the researcher and nurses, and for the group to which each subject will belong to be disclosed to the researcher only after the participant has been included in the study by a person other than the researcher who has no direct role in the study. To prevent performance bias, nurses who met the inclusion criteria and provided informed consent were assigned to the study and control groups by an independent person according to the randomization list. This ensured the researcher's blinding. Since the researcher provided the training to the intervention group according to the guidelines, blinding of the practitioner was not possible. All participating nurses we
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Individualized developmental care-based group care will be provided to infants according to the guidelines.
  Interventions: Behavioral: Infants will receive group care based on individualized developmental care according to the guide.
- Control group (Active Comparator): Infants will receive routine care.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Infants will receive group care based on individualized developmental care according to the guide. — A guide to implementing group care based on individualized developmental care will be developed, and nurses working in the NICU will be trained in group care practices and how to use the guide.
  Other Names: Care based on guidelines
  Arms: Experimental
Behavioral: Standard care — Nurses working in the NICU will continue to provide standard care. After the study is completed, nurses in the control group will also receive the same training as the other group.
  Arms: Control group

SUMMARY:
The Individualized Developmental Care (IDC) model was developed to minimize the negative impact of the neonatal intensive care environment and to support infants' physiological stability. It supports the practice of clustered care, which refers to grouping routine medical and nursing procedures into a single care time period to reduce handling and allow the infant uninterrupted rest and maintenance of the sleep-wake cycle.

This study aims to develop a clustered care practice guideline and evaluate its effectiveness. The study was designed as a single-blind randomized controlled trial, where the participating nurses will not be informed about their group allocation (intervention or control) to reduce bias.The study will be conducted between July and September 2025 in the level 2 and 3 NICUs of Necmettin Erbakan University Faculty of Medicine Hospital in Konya, Turkey.

The study population includes all 44 nurses working in these NICUs who meet the inclusion criteria and agree to participate. Since the entire population is accessible, total population sampling will be used. After data collection is completed, a post hoc power analysis will be conducted using G*Power (v3.1.9.2).

Data will be collected using the "Descriptive Information Form for the Infant and the Nurse" and the "Clustered Care Practice Guideline". Pre-test data will be collected before training, and post-test data will be collected 4-6 weeks after the training.

The intervention group will receive the Clustered Care Practice Training Based on Individualized Developmental Care in two in-person sessions (approx. 45 minutes per session), delivered in small groups (11-12 participants). A training booklet prepared by the researchers will be distributed at the end of the sessions.

The normality of the data will be assessed using the Kolmogorov-Smirnov test, normal distribution curves, and skewness-kurtosis values. Parametric tests will be used for normally distributed data; non-parametric tests will be used otherwise. A significance level of P<0.05 will be applied.

Ethical approval was obtained from the Ethics Committee of KTO Karatay University Pharmaceutical and Medical Research (decision no: 2022/014, date: 21.06.2022). Institutional permission was obtained from NEU Faculty of Medicine Hospital. Written informed consent will be obtained from all participating nurses and from parents of the observed infants.

DETAILED DESCRIPTION:
Premature infants require intensive care during the early stages of life due to their physiological immaturity and heightened sensitivity to environmental stimuli. Routine care practices commonly performed in neonatal intensive care units (NICUs) may negatively affect the comfort and physiological stability of these infants. Therefore, individualized and developmentally supportive care practices tailored to the specific needs of premature infants have become essential.

This randomized controlled trial aims to evaluate the effectiveness of a clustered care practice guideline developed in accordance with individualized developmental care principles. The study will be conducted with nurses working in a neonatal intensive care unit. Nurses will be randomly assigned to either an intervention group or a control group.

The intervention group will receive training on the use of a clinical guideline designed to implement clustered care based on individualized developmental care, while the control group will continue to provide standard routine care. The effectiveness of the intervention will be assessed through the average scores obtained from the use of the guideline and a qualitative analysis of nurses' perspectives. This study is expected to highlight the importance of developmental care approaches in nursing and contribute to enhancing the overall quality of care provided in NICUs.

ELIGIBILITY:
Inclusion Criteria:

* Working in the NICU of Necmettin Erbakan University Medical Faculty Hospital,

  * Having at least 3 months of experience in the NICU,
  * Volunteering to participate in the research.

Exclusion Criteria:

* The nurse wanting to leave the study during the study

  * The nurse not participating in the training or not completing the training
  * The nurse not being able to complete the study, including the final

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Nurse behavior change | within 6 weeks
  Measured by test score change from pre- to post-test within 6 weeks

SECONDARY OUTCOMES:
Nurses' opinions on the effectiveness of the clinical guideline | 4-6 weeks post-intervention
  Evaluation of nurses' perceptions regarding the effectiveness, applicability, and usability of the individualized developmental clustered care guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Geçkil, MD, PhD, Study Director — Necmettin Erbakan University
Locations (1):
- Meram Faculty of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Confidentiality